CLINICAL TRIAL: NCT03518359
Title: Enhanced Resilience Training to Improve Mental Health, Stress and Performance in Resident Physicians
Brief Title: Enhanced Stress Resilience Training for Residents
Acronym: ESRT-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-24601
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Stress; Mindfulness; Cognitive Change
Keywords: Residents; Stress; Well-being

STUDY DESIGN:
Intervention Model Description: Randomized, partially-blinded.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not know that the investigator is testing mindfulness. Participants only will be told that they will be learning stress-reduction skills for physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Training for Residents (Experimental): The intervention will be the modified form of Mindfulness-Based Stress Reduction (MBSR). For this study investigator named the experimental arm Enhanced Stress Resilience Training (ESRT).
  Interventions: Behavioral: Enhanced Stress Resilience Training (ESRT)
- Active Control (Active Comparator): Active control that emphasizes externalized attention via the "shared reading and listening" model.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Enhanced Stress Resilience Training (ESRT) — ESRT involves six weekly 90-minute group classes and one 2 - 4 hour retreat. Classes focus on developing mindfulness skills (i.e. sustained attention, open monitoring, emotional regulation, meta-cognition) in the context of skills and concepts for managing stress, particularly in practicing medicine. Homework consists of 20 minutes per day of mindfulness exercises following guided meditation CDs or videos of movement-based practice, and practice will be reported periodically by text. A 3-hour outdoor retreat occurs at week six. The central exercises of ESRT are the body scan, sitting meditation, chi gong and yoga. For both arms, the weekly teaching sessions occur on a workday morning during protected time at Parnassus, Mission Bay or Zuckerberg San Francisco General Hospital campus.
  Other Names: Modified MBSR
  Arms: Mental Training for Residents
Behavioral: Active Control — Control group participants will meet for 6 weeks, 90 minutes each week, for classes focuses on stress management through rest and exercise, with equivalent protected time and small group bonding but without the use of contemplative practices. Topics will include the history of surgery, patient perspective, the physician personality, technical mastery, fallibility and limits, balancing compassion and detachment and knowing when not to operate. For daily practice, control participants will be asked to devote 20 min per day to stress management through rest and exercise again reported daily by text.
  Arms: Active Control

SUMMARY:
Burnout and overwhelming stress are growing issues in medicine and are associated with mental illness, performance deficits and diminished patient care. Among surgical trainees, high dispositional mindfulness decreases these risks by 75% or more, and formal mindfulness training has been shown feasible and acceptable. In other high-stress populations formal mindfulness training has improved well-being, stress, cognition and performance, yet the ability of such training to mitigate stress and burnout across medical specialties, or to affect improvements in the cognition and performance of physicians, remains unknown. To address these gaps and thereby promote the wider adoption of contemplative practices within medical training, investigators have developed Enhanced Stress Resilience Training, a modified form of MBSR - streamlined, tailored and contextualized for physicians and trainees. Investigators propose to test Enhanced Stress Resilience Training (ESRT), versus active control and residency-as-usual, in surgical and non-surgical residents evaluated for well-being, cognition and performance changes at baseline, post-intervention and six-month follow-up.

DETAILED DESCRIPTION:
Experiencing joy in the practice of medicine is by no means guaranteed. For many physicians, the unique bond with patients, the deep satisfaction of saving a life, and a profound sense of calling make the sacrifice and heartache worthwhile. In contrast, the growing prevalence of burnout, and mental distress is being linked to diminished physician performance, patient outcomes, and hospital economics. This suggests that demands are outstripping resources, thereby threatening the physician-patient bond and the societal pillar this represents.

Overwhelming stress without adequate coping skills has been posited to promote burnout and distress, and may promote performance deficits (from surgical errors to poor professionalism) by impairing cognition and self-regulation. In other high-stress/high-performance groups formal mindfulness training has been shown to enhance stress resilience, subjective well-being and performance. Nevertheless, quality research involving physicians, the effects of chronic stress on performance and the impact of mindfulness training in this context remains scarce, contributing to the slow adoption of mindfulness training into medical practice and residency.

To address these gaps, we first laid the groundwork: we conducted a national survey which showed high dispositional mindfulness in surgery residents reduced the risk of burnout and distress by 75% or more. We conducted a RCT of MBSR in surgery interns, demonstrating feasibility and acceptability of formal mindfulness training. Finally, we have developed an MBSR-based, streamlined curriculum tailored for physicians and trainees, Enhanced Stress Resilience Training (ESRT), which has been beta-tested in surgery faculty and mixed-level residents and refined in terms of logistics, dose and delivery. We have since disseminated our promising results, thereby allowing us access to a larger study population for our proposed RCT of ESRT in mixed-specialty interns as a means to improve well-being, cognition and performance.

While this study will likely not reach statistical power, it will absolutely allow for broader vetting of the curriculum, our current data acquisition and management methods, and the appropriateness of our outcome measures, paving the way for a high-quality, fully-powered MCT in the near future.

The significance of studying mindfulness mental training in medical and surgical trainees is two-fold. One, as a process-centered skill with demonstrated effects on psychological well-being, perceived stress, cognitive performance and physiologic health mindfulness presents a potential gateway mechanism for providing individuals with a 'universal tool' for challenges across all stages of medical training and practice. This includes burnout and errors which are looming issues, largely immutable for the last decade. Two, if feasibility and efficacy among medical and surgical trainees can be shown, the social clout of impacting such a high stress and high performance field is uniquely powerful and could further the dissemination of evidence-based mindfulness interventions to a remarkable degree. Finally, the resultant tendency for enhanced self-awareness and equipoise has been contagious in other settings, providing fuel for a greater culture change in medicine that is much-needed and holds great promise for patients and providers.

The innovation of this work is in bringing a mind-body intervention to bear not only on well-being but also on the fundamental cognitive processes believed to sub-serve performance, such as the impact of attention and working memory capacity on medical decision-making, and the impact of emotional regulation and self-awareness on professionalism and team work. The potential to improve both the operative and clinical environments as well as medical errors is unprecedented. Finally, a vetted, manualized curriculum specifically crafted for physicians could accelerate dissemination nationally.

ELIGIBILITY:
Inclusion Criteria:

* Any consented medical intern from Emergency Medecine, Internal Medicine, Pediatrics, Family Practice, OBGYN and Surgery Depratments in-coming to University of California San Francisco in the study year.

Exclusion Criteria:

* Current personal mindfulness practice, once a week or more frequent;
* Use of medications with Central Nervous System effects;
* Lifetime history of an organic mental illness;
* Acute or chronic immune or inflammatory disorders;
* Pregnancy;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in executive function: National Institutes of Health Examiner battery | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Executive function as assessed via working memory capacity, cognitive control and executive composite components of the NIH EXAMINER battery.
  NIH EXAMINER Battery measures working memory, inhibition, set shifting, fluency, planning, insight, and social cognition and behavior. The EXAMINER battery software calculates the executive composite and factor scores in the R language.

SECONDARY OUTCOMES:
Change in psychological well-being: Mental Health Continuum | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Mental Health Continuum Short Version consists of 14 items that were chosen as the most prototypical items representing the construct definition for each facet of well-being. 6-point Likert scale, from Never (0) to Every Day (5).
Change in psychological well-being: Perceived Stress | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Cohen's Perceived Stress Scale: 10-items, 5-point Likert scale, 0-4. Stress is evaluated as continuous variable or as categorical variable, with high stress is score set at >20 for females and >18 for males.
Change in psychological well-being: Burnout | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Burnout: 2-item Maslach Burnout Inventory, 7-point Likert scale, 0 to 6. High burnout present if either question scores ≥4.
Change in psychological well-being: Anxiety | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Spielberger's State Trait Anxiety index, 4-point Likert, 1 to 4. High anxiety > 40.
Change in psychological well-being: Depression | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Depression and Suicidal Ideation are assessed using the 9-item form of the Patient Health Questionnaire. 4-point Likert scale, 0 to 3 and a total score from 0 to 27 is calculated. Severe depression > 20.
Change in psychological well-being: Mindfulness | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Cognitive and Affective Mindfulness Scale-Revised. 4-point Likert scale, 1 to 4. High mindfulness ≥ 31.
Change in psychological well-being: Alcohol Misuse | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  The AUDIT Alcohol Consumption Questions, 5-point Likert scale, 0 to 4. Misuse for females if score ≥ 3, for males if score ≥ 4.

OTHER OUTCOMES:
Functional neuroanatomic changes | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  Functional changes in areas associated with reappraisal/emotional regulation (amygdala, hippocampus, reward circuitry, appraisal pathway) as evidenced by fMRI BOLD and DTI brain scans analyzed by whole brain and a prior region of interest approaches.
Motor skills | Baseline; 6 weeks post-intervention (9-10wk after baseline), 6 months follow-up.
  Performance as assessed by the Fundamentals of Laparoscopic Surgery (FLS) modules
Mind-Wandering | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  The Mind-Wandering Questionnaire, 5 item scale that is measured the frequency of mind-wandering. 6-point Likert scale, 1 to 6. The total is the sum of the five items within a 5-30 range.
Change in Emotional Regulation: Decentering | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  The Experiences Questionnaire is a 12 item instrument that assesses decentering. 5-point Likert scale,1 to 5.
Change in Performance: Consultation and Relational Empathy | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  The Consultation and Relational Empathy Measure is a validated 10-item questionnaire measuring patient perceptions of empathetic behaviors. 5-point Likert scale from "poor (1)" to "excellent (5)". Score is totaled (10-50 points), with higher scores indicating more empathic behavior.
Change in Performance: Patient Experience | Baseline; post-intervention (9-10wk after baseline), 6 months follow-up.
  The Patient Enablement Instrument is a six-item questionnaire measuring enablement, a concept related to patient satisfaction, but more specific to the physician's patient-centeredness and empowerment. 3-point Likert scale of "much better," "better," and "same or less." Score is totaled (0-12 points), with higher scores indicating greater enablement.

CONTACTS AND LOCATIONS:
Overall Officials: Carter K Lebrares, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Scheepers RA, Boerebach BC, Arah OA, Heineman MJ, Lombarts KM. A Systematic Review of the Impact of Physicians' Occupational Well-Being on the Quality of Patient Care. Int J Behav Med. 2015 Dec;22(6):683-98. doi: 10.1007/s12529-015-9473-3. PMID 25733349
- [Background] Haas JS, Cook EF, Puopolo AL, Burstin HR, Cleary PD, Brennan TA. Is the professional satisfaction of general internists associated with patient satisfaction? J Gen Intern Med. 2000 Feb;15(2):122-8. doi: 10.1046/j.1525-1497.2000.02219.x. PMID 10672116
- [Background] DiMatteo MR, Sherbourne CD, Hays RD, Ordway L, Kravitz RL, McGlynn EA, Kaplan S, Rogers WH. Physicians' characteristics influence patients' adherence to medical treatment: results from the Medical Outcomes Study. Health Psychol. 1993 Mar;12(2):93-102. doi: 10.1037/0278-6133.12.2.93. PMID 8500445
- [Background] Del Canale S, Louis DZ, Maio V, Wang X, Rossi G, Hojat M, Gonnella JS. The relationship between physician empathy and disease complications: an empirical study of primary care physicians and their diabetic patients in Parma, Italy. Acad Med. 2012 Sep;87(9):1243-9. doi: 10.1097/ACM.0b013e3182628fbf. PMID 22836852
- [Background] Sinsky CA, Dyrbye LN, West CP, Satele D, Tutty M, Shanafelt TD. Professional Satisfaction and the Career Plans of US Physicians. Mayo Clin Proc. 2017 Nov;92(11):1625-1635. doi: 10.1016/j.mayocp.2017.08.017. Epub 2017 Nov 1. PMID 29101932
- [Background] Dyrbye LN, Trockel M, Frank E, Olson K, Linzer M, Lemaire J, Swensen S, Shanafelt T, Sinsky CA. Development of a Research Agenda to Identify Evidence-Based Strategies to Improve Physician Wellness and Reduce Burnout. Ann Intern Med. 2017 May 16;166(10):743-744. doi: 10.7326/M16-2956. Epub 2017 Apr 18. No abstract available. PMID 28418518
- [Background] Shirley ED, Sanders JO. Patient satisfaction: Implications and predictors of success. J Bone Joint Surg Am. 2013 May 15;95(10):e69. doi: 10.2106/JBJS.L.01048. PMID 23677370
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Campbell J, Prochazka AV, Yamashita T, Gopal R. Predictors of persistent burnout in internal medicine residents: a prospective cohort study. Acad Med. 2010 Oct;85(10):1630-4. doi: 10.1097/ACM.0b013e3181f0c4e7. PMID 20881685
- [Background] Center C, Davis M, Detre T, Ford DE, Hansbrough W, Hendin H, Laszlo J, Litts DA, Mann J, Mansky PA, Michels R, Miles SH, Proujansky R, Reynolds CF 3rd, Silverman MM. Confronting depression and suicide in physicians: a consensus statement. JAMA. 2003 Jun 18;289(23):3161-6. doi: 10.1001/jama.289.23.3161. PMID 12813122
- [Background] Karlamangla AS, Singer BH, McEwen BS, Rowe JW, Seeman TE. Allostatic load as a predictor of functional decline. MacArthur studies of successful aging. J Clin Epidemiol. 2002 Jul;55(7):696-710. doi: 10.1016/s0895-4356(02)00399-2. PMID 12160918
- [Background] Arora S, Sevdalis N, Aggarwal R, Sirimanna P, Darzi A, Kneebone R. Stress impairs psychomotor performance in novice laparoscopic surgeons. Surg Endosc. 2010 Oct;24(10):2588-93. doi: 10.1007/s00464-010-1013-2. Epub 2010 Mar 31. PMID 20354878
- [Background] Wetzel CM, Kneebone RL, Woloshynowych M, Nestel D, Moorthy K, Kidd J, Darzi A. The effects of stress on surgical performance. Am J Surg. 2006 Jan;191(1):5-10. doi: 10.1016/j.amjsurg.2005.08.034. PMID 16399098
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Background] Amutio A, Martinez-Taboada C, Delgado LC, Hermosilla D, Mozaz MJ. Acceptability and Effectiveness of a Long-Term Educational Intervention to Reduce Physicians' Stress-Related Conditions. J Contin Educ Health Prof. 2015 Fall;35(4):255-60. doi: 10.1097/CEH.0000000000000002. PMID 26953856
- [Background] Johnson DC, Thom NJ, Stanley EA, Haase L, Simmons AN, Shih PA, Thompson WK, Potterat EG, Minor TR, Paulus MP. Modifying resilience mechanisms in at-risk individuals: a controlled study of mindfulness training in Marines preparing for deployment. Am J Psychiatry. 2014 Aug;171(8):844-53. doi: 10.1176/appi.ajp.2014.13040502. PMID 24832476
- [Background] Lebares CC, Guvva EV, Ascher NL, O'Sullivan PS, Harris HW, Epel ES. Burnout and Stress Among US Surgery Residents: Psychological Distress and Resilience. J Am Coll Surg. 2018 Jan;226(1):80-90. doi: 10.1016/j.jamcollsurg.2017.10.010. Epub 2017 Oct 26. PMID 29107117
- [Background] Wager TD, Davidson ML, Hughes BL, Lindquist MA, Ochsner KN. Prefrontal-subcortical pathways mediating successful emotion regulation. Neuron. 2008 Sep 25;59(6):1037-50. doi: 10.1016/j.neuron.2008.09.006. PMID 18817740
- [Result] Lebares CC, Guvva EV, Olaru M, Sugrue LP, Staffaroni AM, Delucchi KL, Kramer JH, Ascher NL, Harris HW. Efficacy of Mindfulness-Based Cognitive Training in Surgery: Additional Analysis of the Mindful Surgeon Pilot Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e194108. doi: 10.1001/jamanetworkopen.2019.4108. PMID 31125095
- [Derived] Lebares CC, Coaston TN, Delucchi KL, Guvva EV, Shen WT, Staffaroni AM, Kramer JH, Epel ES, Hecht FM, Ascher NL, Harris HW, Cole SW. Enhanced Stress Resilience Training in Surgeons: Iterative Adaptation and Biopsychosocial Effects in 2 Small Randomized Trials. Ann Surg. 2021 Mar 1;273(3):424-432. doi: 10.1097/SLA.0000000000004145. PMID 32773637
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860